CLINICAL TRIAL: NCT03168932
Title: Detecting and Quantifying Sulci and White Matter in Fetus' Brain Along the Third Stage of Gestation
Brief Title: Quantification of Fetal Brains' Sulci Along Gestation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yuval Ginsberg, MD, Principal investigator, Rambam Health Care Campus
Other Study IDs: 0398-14-RMB
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Fetal Brain Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gyrogenesis is an ontogenic process that transforms the smooth (lissencephalic) cortex toward its mature, convolved (gyrencephalic) state. A tortuous, branching and deepening pattern of sulci and fissures outlines for a well-developed cortex.

The aim of this study is to find an algorithm that can detect the sulci in ultrasound images of fetus' brain and measure the length of it. This algorithm can be used for research demands like learning the development of the brain from embryo stages until the birth of the baby

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-35
* Gestational age between 25-40 weeks
* Low risk pregnancies

Exclusion Criteria:

* Multiple gestation
* Fetal brain abnormality

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy pregnant women between the age of 18-35 at gestational age of 25-40 weeks
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
morphological changes of the developing fetal brain | 9 months
  Ultrasound measurements of the fetal brain sulcation by a computerized algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided